CLINICAL TRIAL: NCT01362634
Title: A Self-Assessment Intervention for Young Adult Polydrug Users at Risk for HIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Steven Kurtz, Ph.D., Professor, Nova Southeastern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 7R01DA019048 (NIH)
Record Dates: First submitted 2011-05-26; First posted 2011-05-30 (Estimated); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: HIV Infection; Substance Abuse
Keywords: HIV/AIDS; substance use; club drugs; sexual risk
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CAPI Intervention (Experimental): an interviewer-administered comprehensive health and social risk assessment intervention
  Interventions: Behavioral: Trans-theoretical Process of Change Model - interviewer
- ACASI Intervention (Experimental): self-administered comprehensive health and social risk assessment intervention
  Interventions: Behavioral: Trans-theoretical Process of Change Model-self
- Control (No Intervention): waitlist control condition

INTERVENTIONS:
Behavioral: Trans-theoretical Process of Change Model-self — self-administered, computer-based intervention
  Arms: ACASI Intervention
Behavioral: Trans-theoretical Process of Change Model - interviewer — interviewer-administered intervention
  Arms: CAPI Intervention

SUMMARY:
The proposed study is a three-armed randomized clinical trial. A total of 750 clients will be randomly assigned (using a random number table) to the interviewer-administered intervention, the self-administered intervention, and waitlist control conditions upon completion of screening, informed consent, HIV pretest counseling and test administration, and collection of baseline risk behavior data. Outcomes will be measured at 3, 6 and 12 months.

DETAILED DESCRIPTION:
The specific aims of the 5-year study are to:

1. identify the covariates of baseline substance abuse and sexual risks (including demographics, social risk measures, peer norms, abuse history, and mental health status) among a sample of 750 heterosexually active, not-in-treatment, club and prescription drug users ages 18 to 39 in Miami, Florida.
2. evaluate, through random assignment, the relative effectiveness of two intervention conditions and a waitlist control in reducing sex risks and drug use, as measured at 3-, 6- and 12-month follow-ups:

   * Arm 1, an interviewer-administered comprehensive health and social risk assessment intervention (CAPI Intervention) similar to the baseline instrument used in the parent grant;
   * Arm 2, an identical self-administered comprehensive assessment intervention (ACASI Intervention); and
   * Arm 3, a waitlist control condition (Control). Outcome measures, including past 90-day counts of unprotected sex acts and days' drug use, will be obtained from brief risk behavior inventories at baseline and follow-ups.
3. conduct qualitative process evaluation research with 40 participants in each study arm to contextualize the study findings and intervention outcomes.

ELIGIBILITY:
Inclusion Criteria:

* heterosexually active
* ongoing club and prescription drug use
* between 18-39 years of age
* must go to local clubs at least two times per month

Exclusion Criteria:

* no current working phone number or e-mail address
* no intention to remain in South Florida for the next 12 months
* new HIV diagnosis in the past 90 days
* currently participating in a drug treatment program (excluding 12-step programs such as Alcoholics Anonymous)

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 750 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
unprotected sexual intercourse events outside of primary relationships | 3 months
unprotected sexual intercourse events outside of primary relationship | 6 months
unprotected sexual intercourse events outside of primary relationship | 12 months
Days drug use in the past 90 days | 3 months
Days drug use in the past 90 days | 6 months
Days drug use in the past 90 days | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- NSU Research Center, Miami, Florida, United States